CLINICAL TRIAL: NCT00625950
Title: Effect of Treatment With Agonist Dopaminergics on Endometriosic Lesions.
Brief Title: Endometriosis Patients Undergoing Quinagolide Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Prof. Dr. Antonio Pellicer, Instituto Valenciano de Infertilidad, Spain
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VLC-AP-10208-208-1
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Hyperprolactinemia; Endometriosis
Keywords: Hyperprolactinemia; Endometriosis; laparoscopy; angiogenesis, VEGF
MeSH Terms: conditions — Hyperprolactinemia; Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ENDOMETRIAL BIOPSY — Two routine laparoscopies in period of three months with endometrial biopsy comparative study performed.

SUMMARY:
Dopamine agonists, such as quinagolide, are able to act on the VEGFR-2 blocking antibodies, diminishing Vascular Endothelial Growth Factor effect on angiogenesis in human endometriotic lesions.

ELIGIBILITY:
Inclusion Criteria:

* Hyperprolactinemia
* Unexplained infertility
* Endometriosis

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
observation of three month treatment with Quinagolida in endometriosis patients | onset and three months after onset

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Valenciano de Infertilidad, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Gomez R, Abad A, Delgado F, Tamarit S, Simon C, Pellicer A. Effects of hyperprolactinemia treatment with the dopamine agonist quinagolide on endometriotic lesions in patients with endometriosis-associated hyperprolactinemia. Fertil Steril. 2011 Mar 1;95(3):882-8.e1. doi: 10.1016/j.fertnstert.2010.10.024. Epub 2010 Nov 5. PMID 21055747